CLINICAL TRIAL: NCT00099593
Title: Phase II Evaluation of Immunization Against Tumor Cells in Subjects With Sezary Syndrome Using Autologous Mature Dendritic Cells
Brief Title: Immunization Against Tumor Cells in Sezary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-002545-01; FD-R-002545-01
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2006-12

CONDITIONS: Cutaneous T-cell Lymphoma; Sezary Syndrome
Keywords: Cutaneous T-cell lymphoma (CTCL); Sezary Syndrome; Mycosis Fungoides; Vaccine
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides

INTERVENTIONS:
Biological: Autologous Dendritic Cell Vaccine

SUMMARY:
This research is being done to look at the safety and value of a vaccine for a cancer found in the blood and skin known as Cutaneous T-cell lymphoma (CTCL) and Sezary Syndrome.

In the laboratory, researches found that special white blood cells, called dendritic cells (DCs), are able to stimulate the immune system (groups of cells that protect the body from germs and diseases) in a way that helps your body fight cancer. Autologous (from your own body) DCs will be prepared (mixed together) in the laboratory with your cancer cell (Sezary cells) to allow your DCs to pick up parts of your Sezary cells to make the vaccine for you.

DETAILED DESCRIPTION:
Although the etiology of CTCL is not completely understood, immunologic factors appear to play an important role.

Dendritic Cell (DC)-tumor cell vaccines have several features that suggest applications for the immunotherapy of human tumors. Importantly, DC-tumor cell immunization has the potential to simultaneously stimulate CD4+ and CD8+ T cell-mediated immunity against multiple tumor antigens.

The vaccine will be prepared from the subject's own blood, obtained during leukapheresis. From leukapheresed blood, monocyte-derived DCs and malignant lymphocytes will be isolated. The DCs will then be loaded with lymphocyte-derived tumor antigens. Formulations and release criteria must be met before vaccine can be administered.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Sezary syndrome
* Must be willing to discontinue concomitant medications for CTCL, including: *Oral steroids above 10 mg - 30 day washout, unless subject has Addison's Disease or adrenal insufficiency, *PUVA or UVB - 2 week washout, sunbathing, tanning beds, etc. and for the duration of the study, *Electron Beam - for the duration of the study, *Chemotherapeutic agents - 30 day washout, *Bexarotene capsules or other oral biologics - 3 week washout, *Topical nitrogen mustard - 2 week washout, *Extracorporeal photopheresis - 4 week washout and for the duration of the study.
* Must be at least 18 years of age and must be able to understand the written informed consent.
* Subjects must have no evidence of active infection. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible for continuation of therapy after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.

Exclusion Criteria:

* Subjects with autoimmune disease, HIV, and/or hepatitis
* Subjects who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2004-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Clinical response (clearance of skin lesions, clinical and radiographic improvement in lymphadenopathy)

SECONDARY OUTCOMES:
Biological response
Survival
Activities of daily living
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J. Geskin, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Department of Dermatology, Pittsburgh, Pennsylvania, United States